CLINICAL TRIAL: NCT03126448
Title: Prospective Evaluation of Bacterial Burden in Orthopaedic Trauma Procedures Using Highly Sensitive Assays
Brief Title: BBOT: Bacterial Burden in Ortho Trauma Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert O'Toole, Head of the UM SOM's Division of Orthopaedic Traumatology and Chief of Orthopaedics for the University of Maryland Medical Center's (UMMC) R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HP-00066769
Record Dates: First submitted 2017-04-18; First posted 2017-04-24 (Actual); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Orthopaedic Trauma Infections
Keywords: Infection; Nonunion; Fracture healing
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Closed Index Fractures (Other): Group 1 is clean, closed fractures undergoing index open reduction internal fixation (ORIF), intramedullary nailing (IMN) where the fracture site is accessible, or staged treatment of a pilon or plateau that was initially treated by joint spanning external fixation. Tissue obtained at the time of surgery will be sent to the research laboratory for culture and performance of the two highly sensitive assays.
  Interventions: Diagnostic Test: Highly Sensitive Assays
- Group 2: Hardware Removal from Healed Fractures (Other): Group 2 will include patients having a plate removed from a healed fracture without clinical evidence of infection and excluding history of open fracture. Tissue obtained at the time of surgery will be sent to the research laboratory for culture and performance of the two highly sensitive assays.
  Interventions: Diagnostic Test: Highly Sensitive Assays
- Group 3: Index Treatment of Fracture Nonunions (Other): Group 3 will be patients that are undergoing an index procedure for fracture nonunion at a site where prior surgery has been undertaken for the fracture. Exclusions include bone grafting of 'critical' defects, active clinical infection, or < 3 months from index fracture fixation. Tissue obtained at the time of surgery will be sent to the research laboratory for culture and performance of the two highly sensitive assays.
  Interventions: Diagnostic Test: Highly Sensitive Assays

INTERVENTIONS:
Diagnostic Test: Highly Sensitive Assays — Tissue will be collected at the time of surgery from patients in each arm of the study. In addition to tissue stored in RNAlater and sent to a research laboratory, cultures will also be sent to Quest Diagnostics for independent culture results.
  Other Names: Ibis T5000 biosensor; Illumina MiSeq system

SUMMARY:
The purpose of this research project is to improve understanding of the potential role of highly sensitive bacterial tests in diagnosing infected non-healing fractures compared to the current standard of care, microbiologic culture (growing bacteria from tissue specimens in the laboratory).

In order to understand the validity of the highly sensitive tests, parameters of the test in different groups of patients must be established. This study is examining how two highly sensitive tests compare to each other and to the standard of care (microbiologic culture) in three groups of patients.

Group 1 is clean broken bone surgery undergoing plate and screw fixation, intramedullary nailing fixation where the fracture site is accessible, or staged treatment of a broken bones initially treated by joint spanning external fixation device. Group 2 will include patients having a plate and screws removed without clinical evidence of infection. Group 3 will be patients undergoing an initial procedure for fracture nonunion.

DETAILED DESCRIPTION:
Infected, broken bones that do not heal are a difficult clinical problem that significantly affect patient quality of life. Current methodology for detecting bacteria (growth in laboratory cultures) is inadequate to detect infections caused by bacteria existing in a biofilm, which is the layer of "slime" found in the presence of foreign bodies (eg, implanted metal devices to fix broken bones). Advances in molecular biology have allowed development of highly sensitive tests to detect bacteria in the biofilm state. However, the limited prior research has not included control groups or compared the performance of different highly sensitive tests. To address these limitations and further define the role of highly sensitive bacterial tests in clinical practice, the investigators hypothesize that there will be increasing bacterial burden when comparing clean broken bone surgery (1st surgery) to implanted metal device removal (2nd surgery, bone healed) to index nonunion surgery (subsequent surgery, bone not healed) as measured by percentage of cases being positive for bacteria using highly sensitive bacterial tests. Further, the highly sensitive bacterial tests (Illumina MiSeq system and Ibis T5000 biosensor) will have similar ability to quantify the number of bacteria and differentiate bacterial species. Eligible patients will consist of three groups. Group 1 is clean broken bone surgery undergoing plate and screw fixation, intramedullary nailing fixation where the fracture site is accessible, or staged treatment of a broken bones initially treated by joint spanning external fixation device. Group 2 will include patients having a plate and screws removed without clinical evidence of infection. Group 3 will be patients undergoing an initial procedure for fracture nonunion. Tissue obtained at the time of surgery will be sent to the research laboratory for culture and performance of the two highly sensitive tests. The tissue samples taken will be tissue normally removed and discarded in the course of these particular procedures. The rates of positivity for culture and the highly sensitive tests will be compared amongst the three groups. Investigators will also compare bacterial count and the distribution of bacterial species found using the two highly sensitive tests. These data will then undergo statistical analysis against clinical data gathered from review of the patients' charts. The overall project goal is to establish the clinical relevance of highly sensitive bacterial tests in diagnosing infected nonunions. The ability to more accurately identify patients with infection may lead to a change in clinical decision making with respect to surgical procedure or antibiotic treatment. This project will develop an improved understanding of the potential role of highly sensitive bacterial tests in diagnosing infected nonunions compared to the current standard of care, which is growing bacteria in the laboratory under artificial conditions.

ELIGIBILITY:
Inclusion Criteria:

* Closed fracture undergoing open reduction internal fixation, intramedullary nailing (IMN) where the fracture site is accessible, or staged treatment of a pilon or plateau that was initially treated by joint spanning external fixation.
* Plate and screw removal without clinical evidence of infection
* Index procedure for fracture nonunion

Exclusion Criteria:

* Index fracture surgery for an open fracture or intramedullary nailing with fracture site not accessible
* Hardware removal if fracture not already healed
* Index nonunion surgery being bone grafting of a 'critical' defect
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert V O'Toole, MD, Principal Investigator — University of Maryland, College Park; Mark Shirtliff, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Shock Trauma Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Palmer MP, Altman DT, Altman GT, Sewecke JJ, Ehrlich GD, Hu FZ, Nistico L, Melton-Kreft R, Gause TM 3rd, Costerton JW. Can we trust intraoperative culture results in nonunions? J Orthop Trauma. 2014 Jul;28(7):384-90. doi: 10.1097/BOT.0000000000000043. PMID 24343249
- [Background] Stucken C, Olszewski DC, Creevy WR, Murakami AM, Tornetta P. Preoperative diagnosis of infection in patients with nonunions. J Bone Joint Surg Am. 2013 Aug 7;95(15):1409-12. doi: 10.2106/JBJS.L.01034. PMID 23925746
- [Background] Bose D, Kugan R, Stubbs D, McNally M. Management of infected nonunion of the long bones by a multidisciplinary team. Bone Joint J. 2015 Jun;97-B(6):814-7. doi: 10.1302/0301-620X.97B6.33276. PMID 26033062
- [Background] Olszewski D, Streubel PN, Stucken C, Ricci WM, Hoffmann MF, Jones CB, Sietsema DL, Tornetta P 3rd. Fate of Patients With a "Surprise" Positive Culture After Nonunion Surgery. J Orthop Trauma. 2016 Jan;30(1):e19-23. doi: 10.1097/BOT.0000000000000417. PMID 26270457
- [Background] Schottel PC, O'Connor DP, Brinker MR. Time Trade-Off as a Measure of Health-Related Quality of Life: Long Bone Nonunions Have a Devastating Impact. J Bone Joint Surg Am. 2015 Sep 2;97(17):1406-10. doi: 10.2106/JBJS.N.01090. PMID 26333735
- [Background] Brinker MR, Hanus BD, Sen M, O'Connor DP. The devastating effects of tibial nonunion on health-related quality of life. J Bone Joint Surg Am. 2013 Dec 18;95(24):2170-6. doi: 10.2106/JBJS.L.00803. PMID 24352770
- [Background] Hannigan GD, Hodkinson BP, McGinnis K, Tyldsley AS, Anari JB, Horan AD, Grice EA, Mehta S. Culture-independent pilot study of microbiota colonizing open fractures and association with severity, mechanism, location, and complication from presentation to early outpatient follow-up. J Orthop Res. 2014 Apr;32(4):597-605. doi: 10.1002/jor.22578. Epub 2014 Jan 3. PMID 24395335
- [Background] Moussa FW, Anglen JO, Gehrke JC, Christensen G, Simpson WA. The significance of positive cultures from orthopedic fixation devices in the absence of clinical infection. Am J Orthop (Belle Mead NJ). 1997 Sep;26(9):617-20. PMID 9316724
- [Background] Dobbins JJ, Seligson D, Raff MJ. Bacterial colonization of orthopedic fixation devices in the absence of clinical infection. J Infect Dis. 1988 Jul;158(1):203-5. doi: 10.1093/infdis/158.1.203. No abstract available. PMID 3392414
- [Background] Jacovides CL, Kreft R, Adeli B, Hozack B, Ehrlich GD, Parvizi J. Successful identification of pathogens by polymerase chain reaction (PCR)-based electron spray ionization time-of-flight mass spectrometry (ESI-TOF-MS) in culture-negative periprosthetic joint infection. J Bone Joint Surg Am. 2012 Dec 19;94(24):2247-54. doi: 10.2106/JBJS.L.00210. PMID 23318615
- [Background] Struijs PA, Poolman RW, Bhandari M. Infected nonunion of the long bones. J Orthop Trauma. 2007 Aug;21(7):507-11. doi: 10.1097/BOT.0b013e31812e5578. PMID 17762489
- [Background] Motsitsi NS. Management of infected nonunion of long bones: the last decade (1996-2006). Injury. 2008 Feb;39(2):155-60. doi: 10.1016/j.injury.2007.08.032. Epub 2008 Jan 29. PMID 18234202
- [Background] Firoozabadi R, Alton T, Wenke J. Novel Strategies for the Diagnosis of Posttraumatic Infections in Orthopaedic Trauma Patients. J Am Acad Orthop Surg. 2015 Jul;23(7):443-51. doi: 10.5435/JAAOS-D-14-00174. Epub 2015 Jun 3. PMID 26040954
- [Background] Costerton JW, Post JC, Ehrlich GD, Hu FZ, Kreft R, Nistico L, Kathju S, Stoodley P, Hall-Stoodley L, Maale G, James G, Sotereanos N, DeMeo P. New methods for the detection of orthopedic and other biofilm infections. FEMS Immunol Med Microbiol. 2011 Mar;61(2):133-40. doi: 10.1111/j.1574-695X.2010.00766.x. Epub 2011 Jan 18. PMID 21204998
- [Background] Costerton JW. Biofilm theory can guide the treatment of device-related orthopaedic infections. Clin Orthop Relat Res. 2005 Aug;(437):7-11. doi: 10.1097/00003086-200508000-00003. PMID 16056019
- [Background] Dietz FR, Koontz FP, Found EM, Marsh JL. The importance of positive bacterial cultures of specimens obtained during clean orthopaedic operations. J Bone Joint Surg Am. 1991 Sep;73(8):1200-7. PMID 1890121
- [Background] Panousis K, Grigoris P, Butcher I, Rana B, Reilly JH, Hamblen DL. Poor predictive value of broad-range PCR for the detection of arthroplasty infection in 92 cases. Acta Orthop. 2005 Jun;76(3):341-6. PMID 16156461
- [Background] Simpson AH, Wood MK, Athanasou NA. Histological assessment of the presence or absence of infection in fracture non-union. Injury. 2002 Mar;33(2):151-5. doi: 10.1016/s0020-1383(01)00078-x. PMID 11890917
- [Background] ELEK SD. Experimental staphylococcal infections in the skin of man. Ann N Y Acad Sci. 1956 Aug 31;65(3):85-90. doi: 10.1111/j.1749-6632.1956.tb36626.x. No abstract available. PMID 13363202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Closed Index Fractures | Group 2: Hardware Removal From Healed Fractures | Group 3: Index Treatment of Fracture Nonunions
Started | 56 | 49 | 37
Completed | 43 | 41 | 27
Not Completed | 13 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Closed Index Fractures | Group 2: Hardware Removal From Healed Fractures | Group 3: Index Treatment of Fracture Nonunions | Total
Number analyzed (Participants) | 43 | 41 | 27 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (19) | 46 (15) | 47 (14) | 45 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 10 | 50
  Male | 24 | 20 | 17 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 29 | 31 | 21 | 81
ASA Physical Status Classification System [Mean (Standard Deviation); unit: units on a scale] — ASA 1: Healthy Patients
  ASA 2: Mild to moderate systemic disease caused by the surgical condition or by other pathological processes, and medically well controlled
  ASA 3: Severe disease process which limits activity but is not incapacitating
  ASA 4: Severe incapacitating disease process that is a constant threat to life
  ASA 5: Moribund patient not expected to survive 24 hours with or without an operation
  ASA 6: Declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2.1 (0.7) | 2.0 (0.8) | 2.2 (0.5) | 2.1 (0.8)
High Energy Injury [Count of Participants; unit: Participants] | 32 | 32 | 17 | 81
Compartment Syndrome [Count of Participants; unit: Participants] | 0 | 1 | 2 | 3
Pre-operative Antibiotics Administered [Count of Participants; unit: Participants] | 43 | 40 | 26 | 109
Open Fracture [Count of Participants; unit: Participants] | NA — Inclusion criteria or study protocol precluded obtaining this information for acute fractures | 4 | 18 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tissue Samples Identified With Bacterial DNA According to Highly Sensitive Bacterial Assays
Description: The objective of this research is to see if highly sensitive bacterial assays are useful for determining whether fracture nonunions are infected
Time Frame: Study surgery to 6-month clinical follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Closed Index Fractures | Group 2: Hardware Removal From Healed Fractures | Group 3: Index Treatment of Fracture Nonunions
Number analyzed (Participants) | 43 | 41 | 27
Participants | 10 | 24 | 20

ADVERSE EVENTS:
Time Frame: Study enrollment through 6-month follow-up
Arm/Group | Group 1: Closed Index Fractures | Group 2: Hardware Removal From Healed Fractures | Group 3: Index Treatment of Fracture Nonunions
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/41 | 1/27
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/27
Other Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/27

LIMITATIONS AND CAVEATS:
1. Subjective assessment of active infection and fracture union/nonunion by the attending surgeon.
2. Groups were heterogeneous in surgical sites
3. Differential inclusion of open fractures
4. Loss to follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT03126448/Prot_SAP_000.pdf